CLINICAL TRIAL: NCT01103583
Title: Hydroxyurea in Primary Progressive Multiple Sclerosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No efficacy (interim.analysis)
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Marco Salvetti, CENTERS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-008521-29
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyurea (Experimental)
  Interventions: Drug: Hydroxyurea
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Hydroxyurea — 500 mg/die per os for two years
  Arms: Hydroxyurea
Other: placebo — 500 mg/die per os for two years
  Arms: Placebo

SUMMARY:
The pathogenesis of MS remain elusive, however some studies have linked the disease with infection by Epstein-Barr virus; therefore the use of drugs with immunosuppressive or immunomodulating action alone may be less suitable for primary progressive MS.This study will evaluate treatment with hydroxyurea (HU) in primary progressive MS. Hydroxyurea act by inhibiting the synthesis of deoxynucleotides essential for viral transcription,HU has recently been used in combination with antiretroviral drugs in HIV and has been shown to limit immune activation and suppress viral load by both antiviral and cytostatic activities. Furthermore has been demonstrated experimentally that HU suppressed the expression of EBV. For these reasons HU could be useful in primary progressive MS with cytostatic and antiviral action , confirming the role of EBV in the pathogenesis of MS.

ELIGIBILITY:
Inclusion Criteria:

* sign written informed consent
* 18 to 60 years of age inclusive
* diagnosis of PP-MS according to McDonald criteria
* EDSS score at screening of 2-7 inclusive

Exclusion Criteria:

* hypersensitivity to hydroxyurea
* patients who were treated with immunosuppressive drugs or steroid three month before
* respiratory or urinary infections
* history or presence of malignancy
* pregnancy or lactation
* low compliance to the therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
the evaluation of safety and tolerability of hydroxyurea | two years

SECONDARY OUTCOMES:
the evaluation of efficacy of hydroxyurea in primary progressive multiple sclerosis | two yeras

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centre for Experimental Neurological Therapies (CENTERS), Tor Vergata University Hospital, Rome
  - Centre for Experimental Neurological Therapies (CENTERS), S.Andrea Hospital, Rome